CLINICAL TRIAL: NCT06209268
Title: The Impact of Selective Vitamin D Receptor Activation on Clinical Outcomes in Septic Patients -a Randomised Placebo Controlled Trial
Brief Title: The Impact of Selective Vitamin D Receptor Activation on Clinical Outcomes in Septic Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Split, School of Medicine (Other)
Responsible Party: Principal Investigator, Vedran Kovacic, Profesor of Medicine, University of Split, School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: USplitSM111
Record Dates: First submitted 2023-11-21; First posted 2024-01-17 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Sepsis
MeSH Terms: conditions — Sepsis | interventions — paricalcitol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- paricalcitol group (Active Comparator)
  Interventions: Drug: Paricalcitol injection
- placebo group (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Paricalcitol injection — 5 μg intravenous paricalcitol (1 mL) per day in five consecutive days
  Arms: paricalcitol group
Drug: Placebo — 0.9% NaCl 1 ml per day in five consecutive days
  Arms: placebo group

SUMMARY:
Sufficient serum levels of vitamin D are important for immune system regulation with protective effect against severe infection and overactivated inflammatory response in sepsis. It is also not clear what level of vitamin D in the blood would be the trigger for vitamin D administration. A more selective approach to VDR activation than cholecalciferol could have a more significant role in the clinical outcomes of patients with sepsis. A study demonstrated that low baseline serum level of vitamin D receptor (VDR) was associated with a high incidence of 28-day mortality and negatively correlated with lactate, C-reactive protein, APACHE II SOFA scores, and disease severity among patients with sepsis in an ICU setting.

The role of selective vitamin D receptor activation agents (paricalcitol or maxacalcitol) was not studied in septic patients, despite its anti-inflammatory and immunomodulatory properties. Vitamin D analogs have different effects on nuclear VDRs than does calcitriol, through different response elements in various target genes, so it is possible that their effect on a patient with sepsis will be more effective than cholecalciferol. As distribution of VDRs is ubiquitous in many organs and tissues, selective VDR activation with paricalcitol may have beneficial effects in preserving organs functionality and modulating the immune response in sepsis.

Hypotheses

1. The immunoregulatory, anti-inflammatory, and anti-oxidative properties of selective vitamin D receptor activator paricalcitol would result in improvement of inflammatory, endothelial function, and antioxidative parameters and clinical outcomes in groups of septic patient admitted to ICU.
2. The baseline septic patient serum 25(OH) D3 levels at admission time in ICU have influence on clinical outcomes as well as on inflammatory, endothelial function, and antioxidative parameters.
3. The inflammatory, endothelial function, and antioxidative parameters measured at ICU admission time have significant impact on clinical outcomes in septic patients.

The aim

The main objective of study is to test hypothesis that that selective activator of vitamin D receptors paricalcitol will improve outcomes of septic patient admitted in ICU. The study aims to investigate the effects of paricalcitol on clinical outcomes, inflammatory markers, organ dysfunction, endothelial function, vascular morphology, coagulation markers, and haemodynamic parameters.

The additional objectives of the study are to test hypothesis that septic patient serum 25(OH)vitamin D3 have impact on inflammatory, endothelial function, and antioxidative parameters including protein carbonylation; and to test hypothesis that these markers and clinical outcomes are interconnected with significant impact on clinical outcomes.

DETAILED DESCRIPTION:
There are evidences that decreased vitamin D levels among septic patients shown significant associations with adverse outcomes.

The large PETAL-VIOLET trial was conducted in 44 hospitals in the United States and enrolled 1358 severe patients (more than 80% were admitted to the ICU for medical diseases) with vitamin D deficiency. Study protocol included very early vitamin D3 supplementation (a single enteral dose of 540,000 IU) in critically ill. Results showed that early high dose of vitamin D3 supplementation had no advantage over placebo with respect to 90 day mortality or hospital stay, and found no differences between the groups of participants.

Second large study, VITdAL-ICU randomized clinical trial, was conducted among 492 critically ill adult patients with vitamin D deficiency (≤20 ng/mL) assigned to receive either vitamin D3 given orally or via nasogastric tube once at a dose of 540,000 IU followed by monthly maintenance doses of 90,000 IU for 5 months; or a placebo. There was no difference between groups in length of hospital stay, hospital mortality, and 6-month mortality. In severe vitamin D deficiency (≤12 ng/mL) subgroup analysis, only hospital mortality was significantly lower for vitamin D3 receivers.

A recent metaanalysis included 11 randomized control trials with a total of 2187 patients concluded that vitamin D supplementation in critically ill patients decreases the duration of mechanical ventilation and ICU stay. There was no significant difference noted in mortality and length of hospital stay.

Many of these studies on ICU population included mixed ICU population, including also septic patients. Only minority of studies was conducted and dedicated exclusively for septic population. VITdAL-ICU and PETAL-VIOLET trials included critically ill patients with a low prevalence of sepsis at the enrolment time (7.7% and 33.3%), so sepsis subgroup analyses did not allow clear conclusion on the efficacy of vitamin D supplementation in septic patients.

Also, in the future it is necessary to investigate the possible impact of selective activators of vitamin D receptors (for example paricalcitol) among population of patient with sepsis, as it is well known beneficial anti-inflammatory and anti-oxidative properties of paricalcitol on renal and cardiovascular system.

Paricalcitol Several new vitamin D analogues have been developed for treatment of secondary hyperparathyroidisms with a reduced risk of hypercalcemia and hyperphosphatemia. The third generation of vitamin D analogues is composed of a group of 1- and 25-hydroxylated vitamin D compounds with either ring structure modifications (19-nor-1,25-dihydroxyvitamin D2 or paricalcitol). Vitamin D analogues have different effects on nuclear vitamin D receptor than calcitriol, through different response elements in various target genes. Such new vitamin D analogues because of unique properties of nuclear vitamin D receptor are named selective vitamin D receptor activation agents. The term selective means that this molecule acts mostly to parathyroid gland than to intestine and bone, resulting in lower serum calcium and phosphorus blood concentrations. Such selective vitamin D receptor activation agents are reported to have beneficial effects such as anti-inflammatory and antithrombotic effects, inhibition of vascular smooth muscle cell proliferation, inhibition of renin-angiotensin system, inhibition of vascular calcification and stiffening, and regression of left ventricular hypertrophy. Antioxidative properties of paricalcitol are demonstrated in animal model of contrast induced nephropathy as lower levels of serum malondialdehyde and kidney thiobarbituric acid-reacting substances in the paricalcitol group. Paricalcitol was found to decrease angiotensinogen, renin, renin receptor, and vascular endothelial growth factor mRNA levels in rat model of chronic renal failure. In VITAL study, a randomised clinical trial, paricalcitol demonstrated additional lowering effect on albuminuria in patients with diabetic nephropathy. Antifibrotic effects of paricalcitol is demonstrated in animal model that paricalcitol reduces myocardial fibrosis and preserves diastolic left ventricular function due to pressure overload which was associated with a reduced fibrosis. Paricalcitol may prevent the cisplatin-induced kidney injury by suppressing the fibrotic, apoptotic and proliferative factors in animal model; paricalcitol suppressed the expression of TGF-β1, Smad signaling, mitogen-activated protein kinase signaling, p53-induced apoptosis, and p27(kip1).

The aim Effect of selective activation of vitamin D on clinical outcomes in sepsis is completely unknown and there are lack of human studies that would clarify the role of selective activation of receptors for vitamin D in sepsis. Although there is some piece of evidence, which is sometimes controversial, of a beneficial effect of vitamin D on the outcomes of patients with sepsis, a study examined the impact of paricalcitol on septic patients is missing. Therefore, we think that the research of paricalcitol in sepsis is important. Except clinical outcomes, we will included in study markers of inflammation, endothelial function, arterial stiffness and oxidation in aim to provide additional insight into pathophysiological concept of sepsis. It is very important to investigate the possible influence of paricalcitol on some of these markers, and the interrelationship between the markers and the possible favourable clinical impact of paricalcitol on clinical outcomes. Additionally, the second important aim of the study is provide evidence of the association of oxidative, endothelial, inflammatory and other markers with clinical outcomes and with the concentration of vitamin D in the plasma of septic patients.

Participants The participants of this study will be patients admitted as sepsis in a medical ICU. The including criteria for sepsis will be defined according The Third International Consensus Definitions for Sepsis and Septic Shock. The sepsis will be defined as suspected infection with SOFA score>=2. The subgroup of participants with septic shock will be defined as sepsis with vasopressor requirement to maintain a mean arterial pressure of 65 mm Hg or greater and serum lactate level greater than 2 mmol/L despite adequate fluid resuscitation.

Exclusion criteria will be initial total serum calcium ≥2.60 mmol/L, significant chronic end stage heart, kidney or liver disease, active treatment with corticosteroids or cytotoxic drugs, autoimmune diseases, malignancies, and cachexia. Subjects should have not previously been on active vitamin D therapy minimally within the last four months prior to the study period.

All subjects will receive standard care for patients with sepsis according international guidelines for sepsis treatment.

Sample size calculation with confidence level of 90% and margin of error of 10% estimated minimal number of 69 subjects need for the study. We plan to enrolled approximately 40-50 participants in each group of subjects.

Study protocol

All subjects will be randomised (computer generated process) in 1:1 ratio to received placebo or paricalcitol. Enrolment of the subjects will be demonstrated as CONSORT flow diagram.

Intervention phase will last 5 days during ICU staying, whereupon will start follow up phase of trial.

Participants will be randomised to receive 5 μg intravenous paricalcitol (1 mL) per day in five consecutive days, or to receive placebo (1 mL 0.9% NaCl). If serum calcium exceeded 2.65 mmol/L, the intervention will be stopped.

Ethic issues The participants will be informed about the purpose and nature of the study and gave written consent. The study protocol will be accepted by the local University's Hospital Ethics Committee.

Outcome measures

For all subjects will be recorded data on previous diseases, smoking habits, body mass index (BMI) (kg/m2), SOFA score (on 0 and 7 day), SAPS score (on 0 and 7 day), need for RRT, need for mechanical ventilation, classification as sepsis or as septic shock, survival at 7 and 28 days.

Outcome measurements will be performed at baseline, and for some of the outcomes at the seven day of ICU or post-ICU staying. For survival outcome participants will be followed up at 7 and the 28 day.

Clinical outcomes: delta SOFA score (0 and 7 day), delta SAPS score (0 and 7 day), days need for RRT, days need for mechanical ventilation, ICU days stay, survival at 7 and 28 days, days need for catecholamines, admission time MAP, average MAP at day 5 with delta MAP (0 and 5 day), ECG abnormalities during the first 5 days.

Standard laboratory measurements, coagulation and inflammation markers: (at admission time and at day 7): from venous blood specimen: leucocytes count, hemoglobin, plateless count, activated partial thromboplastin time (aPTT), prothrombin time (PT), serum concentration of: urea, creatinine, calcium, phosphorus, albumins, total cholesterol, high-density lipoprotein (HDL)-cholesterol, C-reactive protein (CRP), serum 25(OH)D3, albumins, troponin-I, NT-proB-type natriuretic peptide (NT-proBNP), ferritin, iPTH, fibrinogen, D-dimers, procalcitonin (PCT), bicarbonate, lactate; and blood gasses analysis from arterial specimen. Changes in variables between 0 and 7 days will be recorded.

Oxidative stress: at admission time from venous blood specimen (at admission time): lipid peroxidation products TBARS (ThioBarbituric Acid Reactive Substances) and FOX (Ferrous Oxidation - Xylenol orange assay), and malondialdehyde. Additionally, at admission time from venous blood specimen will be assessed measurement of plasma protein carbonylation as protein carbonyl groups are early markers of protein oxidative damage. The protein carbonyl concentrations will be recorded for all subjects.

Non-invasive assessments of Arterial Stiffness: (at admission time): Applanation tonometry will be used for arterial stiffness assessment. Tonometric transducer will be placed on the carotid and femoral artery to obtain pulse wave velocity (PWV) and for pulse wave analysis (PWA) assessment, a tonometric transducer will be placed on the radial artery. PWA will be consisted from peripheral and central augmentation index (pAIx, cAIx), central pulse pressure (cPP), central systolic and diastolic blood pressure (cSBP, cDBP), central mean blood pressure (cMBP), peripheral pulse pressure (pPP), peripheral systolic and diastolic blood pressure (pSBP, pDBP) and peripheral mean blood pressure (pMBP).

Ultrasonographic studies:

1. Assessment of endothelial function: (at admission time and at day 7): Endothelial function will be determined by recording the dilator response of the brachial artery to increased blood flow generated during reactive hyperaemia of the downstream forearm. Baseline recordings of arterial diameter will be made for one minute before inflation of a blood pressure cuff placed just distal to the elbow. End-diastolic images of the artery were acquired. Reactive hyperaemia will be induced by a pneumatic cuff placed on the forearm distal to the scanned brachial artery, to a pressure of 250 mmHg for 5 min. Analysis of the diameter of brachial artery will be performed at the end of diastole to the rest, 1 min., 2 min., 3. min. and 4 min. after cuff deflation using electronic callipers on the computed system in M-mode of frozen images scanning. Recorded values will be baseline diameter of brachial artery (mm), and differences between baseline deflation diameter, recorded as maximal difference between baseline and diameters after deflation (given as absolute values and as percent of baseline values). Changes in variables between 0 and 7 days will be recorded.
2. Intrarenal arteries spectral analysis: assesment of vascular resistance (at admission time and at day 7): 2D and Doppler ultrasound examination of the both kidneys with estimation of resistance index and pulsatility index (RI and PI) of the intrarenal arterial branches will be measured and recorded as RI and PI mean (left and right kidney). Changes in variables between 0 and 7 days will be recorded.
3. Ultrasound measurement of quadriceps muscle thickness: (at admission time and at day 7): using high-frequency linear probe the muscle thickness of the quadriceps femoral muscle will detected by ultrasound in a transverse scan, including the thickness of the rectus femoris and vastus intermedius. The ultrasound probe will be placed perpendicular to the long axis of the right femur (transverse) on its anterior surface, at the midpoint of the length between the anterior superior iliac spine and the patella. The Quadriceps muscle layer thickness (QMLT) will be provided by measuring the distance between the cortex of the femur and the most superficial muscular fascia by applying maximal compression on the ultrasound probe in order to prevent the reading errors due to subcutaneous edema. Changes in the QMLT between 0 and 7 days will be recorded.
4. ultrasound of the spleen (B-mode) (on admission and on the 7th day): to assess the degree of hardness of the spleen using point shear wave elastography (P-SWE) by repeated measurements of the spleen tissue. The mean value of the degree of hardness (kPa) as well as the degree of attenuation (ATT) (dB/cm/MHz) will be recorded. Finally, the volume of the spleen will be determined. Changes between 0 and 7 days will be recorded.

ELIGIBILITY:
Inclusion Criteria:The participants of this study will be patients:

* admitted as sepsis in a medical ICU. The including criteria for sepsis will be defined according The Third International Consensus Definitions for Sepsis and Septic Shock. The sepsis will be defined as suspected infection with SOFA score>=2.
* The subgroup of participants with septic shock will be defined as sepsis with vasopressor requirement to maintain a mean arterial pressure of 65 mm Hg or greater and serum lactate level greater than 2 mmol/L despite adequate fluid resuscitation.

Exclusion Criteria:

* total serum calcium ≥2.60 mmol/L,
* significant chronic end stage heart, kidney or liver disease
* active treatment with corticosteroids or cytotoxic drugs
* autoimmune diseases
* malignancies
* cachexia
* previously been on active vitamin D therapy the last four months prior to the study period.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2025-10-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
survival (days) | 7. and the 28. day

SECONDARY OUTCOMES:
leucocytes count from venous blood specimen | 0. and the 7. day
  leucocytes count (10 9/L)
blood gasses analysis | 0. and the 7. day
  blood gasses analysis from arterial specimen (PCo2, PO2 in kPa).
Oxidative stress | 7.day
  lipid peroxidation products TBARS (ThioBarbituric Acid Reactive Substances) (μM MDA )and FOX (Ferrous Oxidation - Xylenol orange assay) (μM H2O2.).
Non-invasive assessments of Arterial Stiffness-pulse wave velocity-pulse wave velocity | 0. and the 7. day
  Applanation tonometry will be used for arterial stiffness assessment. Tonometric transducer will be placed on the carotid and femoral artery to obtain pulse wave velocity (PWV) (m/s)
ultrasound of the spleen (B-mode) | 0. and the 7. day
  To assess the degree of hardness of the spleen using point shear wave elastography (P-SWE) by repeated measurements of the spleen tissue. The mean value of the degree of hardness (kPa) as well as the degree of attenuation (ATT) (dB/cm/MHz) will be recorded.
Sequential Organ Failure Assessment (SOFA) | 0., 5. and 7. day
  delta Sequential Organ Failure Assessment (SOFA) score (from 2-24, 0-the best, 15 the worst) (0 and 7 day)
SAPS (Simplified Acute Physiology Score) | 0., 5. and 7. day
  delta SAPS (Simplified Acute Physiology Score) II score (3-163 points, 3 the best, 163 the worst) (0 and 7 day)
days of ICU treatment | 7. day
  days need for renal replacement therapy (RRT) (days) days need for mechanical ventilation (days) ICU (intensive care unit) days stay (days) days need for catecholamines (days)
MAP (mean arterial pressure) | 0., 5. and 7. day
  admission time MAP (mean arterial pressure) (mmHg) average MAP (mean arterial pressure) at day 5 (mmHg) delta MAP (mean arterial pressure) (0 and 5 day) (mmHg)
haematology parameters from venous blood specimen-plateless count | 0. and the 7. day
  plateless (10 9/L) count
coagulation parameters from venous blood specimen- activated partial thromboplastin time | 0. and the 7. day
  activated partial thromboplastin time (aPTT) (sec)
coagulation parameters from venous blood specimen-prothrombin time | 0. and the 7. day
  prothrombin time (PT) (sec)
Non-invasive assessments of Arterial Stiffness-Central Augmentation Index | 0. and the 7. day
  Applanation tonometry will be used for arterial stiffness assessment. Central Augmentation Index is calculated by determining the ratio of Augmentation Pressure (cAP) (mmHg) to Pulse Pressure (cPP) (mmHg): cAIx = cAP / cPP. This is known as the Central Pressure Waveform
Assessment of endothelial function | 0. and the 7. day
  Endothelial function will be determined by recording the dilator response of the brachial artery to increased blood flow generated during reactive hyperaemia of the downstream forearm. Baseline recordings of arterial diameter will be made for one minute before inflation of a blood pressure cuff placed just distal to the elbow. End-diastolic images of the artery were acquired. Reactive hyperaemia will be induced by a pneumatic cuff placed on the forearm distal to the scanned brachial artery, to a pressure of 250 mmHg for 5 min. Analysis of the diameter of brachial artery will be performed at the end of diastole to the rest, 1 min., 2 min., 3. min. and 4 min. after cuff deflation using electronic callipers on the computed system in M-mode of frozen images scanning. Recorded values will be baseline diameter of brachial artery (mm).
Intrarenal arteries spectral analysis: assesment of vascular resistence (RI-resistance index) | 0. and the 7. day
  2D and Doppler ultrasound examination of the both kidneys with estimation of resistance index and pulsatility index (RI and PI) of the intrarenal arterial branches will be measured and recorded as RI and PI mean (left and right kidney).
Ultrasound measurement of quadriceps muscle thickness | 0. and the 7. day
  using high-frequency linear probe the muscle thickness of the quadriceps femoral muscle will detected by ultrasound in a transverse scan, including the thickness of the rectus femoris and vastus intermedius (mm) The ultrasound probe will be placed perpendicular to the long axis of the right femur (transverse) on its anterior surface, at the midpoint of the length between the anterior superior iliac spine and the patella. The Quadriceps muscle layer thickness (QMLT) will be provided by measuring the distance between the cortex of the femur and the most superficial muscular fascia by applying maximal compression on the ultrasound probe in order to prevent the reading errors due to subcutaneous edema.
concentration of creatinin (umol/L) from venous blood specimen | 0. and the 7. day
concentration of calcium (mmol/L)from venous blood specimen | 0. and the 7. day
concentration of phosphorus (mmol/L)from venous blood specimen | 0. and the 7. day
concentration of albumins (g/L)from venous blood specimen | 0. and the 7. day
concentration of total cholesterol (mmol/L)from venous blood specimen | 0. and the 7. day
concentration of high-density lipoprotein (HDL)-cholesterol (mmol/L)from venous blood specimen | 0. and the 7. day
concentration of C-reactive protein (CRP) (mg/L)from venous blood specimen | 0. and the 7. day
concentration of serum 25(OH)D3 (nmol/l)from venous blood specimen | 0. and the 7. day
concentration of troponin-I (mmol/L)from venous blood specimen | 0. and the 7. day
concentration of NT-proB-type natriuretic peptide (NT-proBNP) (mmol/L)from venous blood specimen | 0. and the 7. day
concentration of ferritin (mg/L)from venous blood specimen | 0. and the 7. day
concentration of iPTH (nmol/L)from venous blood specimen | 0. and the 7. day
concentration of fibrinogen (mg/L)from venous blood specimen | 0. and the 7. day
concentration of D-dimers (mg/L)from venous blood specimen | 0. and the 7. day
concentration of procalcitonin (PCT) (mg/mL)from venous blood specimen | 0. and the 7. day
concentration of bicarbonate(mmol/L)from arterial blood specimen | 0. and the 7. day
concentration of lactate (mmol/L)from arterial blood specimen | 0. and the 7. day

CONTACTS AND LOCATIONS:
Overall Officials: Vedran Kovacic, prof.dr., Principal Investigator — University of Split, School of Medicine

IPD SHARING:
Plan to Share IPD: No